CLINICAL TRIAL: NCT06905015
Title: Comparison the Effectiveness of Stroke Volume Variation Versus Central Venous Pressure Guidance for Reducing Perioperative Blood Loss During Open Liver Resection: A Prospective, Double-Blinded, Noninferiority, Randomized Controlled Study
Brief Title: Stroke Volume Variation Versus Central Venous Pressure Guidance for Reducing Perioperative Blood Loss During Open Liver Resection
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Warangkana Lapisatepun (Other)
Collaborators: Chiang Mai University (Other)
Responsible Party: Sponsor-Investigator, Warangkana Lapisatepun, Chiang Mai University, Chiang Mai University
Organization: Chiang Mai University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ANE-2567-0300
Record Dates: First submitted 2025-03-25; First posted 2025-04-01 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Liver Tumor; Surgery; Primary Liver Tumor, Metastatic Liver; Primary Liver Cancer; Liver Resection; Benign Liver Tumor
Keywords: Stroke volume variation; central venous pressure; open liver resection; blood loss
MeSH Terms: conditions — Carcinoma, Hepatocellular; Hemorrhage

STUDY DESIGN:
Intervention Model Description: Noninferiority randomized controlled trials
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High SVV group (Experimental): High stroke volume variation group: Anesthesiologists will perform methods to achieve and maintain SVV at 13-20% during liver parenchymal transection (fluid restrictive phase). Central venous pressure monitoring will be concealed with drapes, and the room anesthesiologist will use SVV for guiding fluid management.
  Interventions: Device: High stroke volume variation group
- Low CVP group (Active Comparator): Low central venous pressure group: Anesthesiologists will perform methods to maintain CVP under 5 mmHg during liver parenchymal transection (fluid restrictive phase). Stroke volume variation monitoring will be concealed by drapes, and the room anesthesiologist will use CVP to guide fluid management.
  Interventions: Device: High stroke volume variation group

INTERVENTIONS:
Device: High stroke volume variation group — Anesthesiologists will perform methods to achieve and maintain SVV at 13-20% during liver parenchymal transection (fluid restrictive phase). Central venous pressure monitoring will be concealed with drapes, and the room anesthesiologist will use SVV for guiding fluid management only during parenchymal transection phase. If SVV exceeds 20%, a balanced salt crystalloid will be administered in the minimal amount necessary to reduce the SVV to below 20%.

SUMMARY:
Liver resection is a major surgery that can be associated with significant intraoperative blood loss and blood transfusion. Among high-volume centers, median intraoperative blood loss ranges between 300-800 ml. Excessive blood loss is a strong independent predictor of worsened postoperative outcomes, increasing morbidity and mortality rates by 20%-35%. Additionally, perioperative allogeneic blood transfusions are associated with deleterious outcomes, including tumor recurrence and increased rates of complications and death.

The liver is a highly vascular organ with minimal vascular resistance, receiving up to 25% of cardiac output and pooling 20% of the splanchnic blood. Hepatic veins are a common source of venous hemorrhage. The pressure in the hepatic veins is directly correlated with the pressure in the vena cava and reducing cardiac preload results in decreased hepatic vein congestion. Therefore, low central venous pressure anesthesia (typically below 5 mmHg) can reduce the pressure gradient for retrograde venous bleeding, facilitate the outflow of blood from hepatic veins, and decrease blood volume and pressure in the liver. This anesthetic method is the standard technique to minimize blood loss during liver resection.

Central venous pressure was the static parameter used to indicate the right ventricular end-diastolic volume index (RVEDI) and was believed to be correlated with volume status. Despite this, central venous pressure did not reliably predict preload responsiveness due to the curvilinear shape of the ventricular pressure-volume curve, which indicates a poor relationship between ventricular filling pressure and volume. Additionally, the placement of a central venous catheter could lead to serious complications such as arterial cannulation, pneumothorax, and infection.

Arterial waveform analysis is dynamic hemodynamic monitoring based on the interaction between the heart and lungs in patients with mechanical ventilation. Stroke volume variation (SVV) is one aspect of arterial pressure waveform analysis and is a less invasive alternative technique for guiding preload status and fluid management in patients undergoing major abdominal surgery.

In liver resection, several anesthetic methods are used to achieve low central venous pressure (CVP < 5 mmHg) during the liver parenchymal dissection phase. These methods include intraoperative volume restriction, administration of venodilators or vasodilators, the use of forced diuresis with furosemide, and the implementation of hypovolemic phlebotomy. As mentioned, central venous pressure is a static hemodynamic monitoring parameter and poorly correlates with volume status. Recently, stroke volume variation has been recognized as a good parameter to predict volume status and fluid responsiveness in patients undergoing liver resection. However, no previous publications have studied the efficacy of stroke volume variation monitoring compared with central venous pressure monitoring to reduce perioperative blood loss during open liver resection.

The study aimed to compare the efficacy of maintaining high stroke volume variation versus low central venous pressure in reducing perioperative blood loss during the liver transection phase in open liver resection.

DETAILED DESCRIPTION:
Bleeding is the most common and concerning complication in liver resection because it affects overall complications. Nowadays, there are numerous surgical and anesthetic techniques to decrease blood loss and the need for blood transfusion during liver resection. Surgical strategies include the use of temporary hepatic vascular occlusion techniques, infrahepatic inferior vena caval clamping, and multiple parenchymal transection techniques to minimize intraoperative blood loss and blood transfusion.

Low central venous pressure (CVP < 5 mmHg) is the main anesthetic technique to reduce blood loss and transfusion requirements. Low CVP decreases the impedance for blood flow through the hepatic venous system into the inferior vena cava, resulting in reduced retrograde venous bleeding during parenchymal resection. Low CVP anesthesia can be achieved by several methods such as restrictive intravenous fluid infusion, administration of diuretics and systemic nitroglycerin, reducing mechanical ventilation, and the application of epidural anesthesia.

Nowadays, stroke volume variation (SVV) monitoring, obtained using the FloTrac-Vigileo system (Edwards Lifesciences®, Irvine, CA, USA), is a minimally invasive technique for hemodynamic monitoring that utilizes arterial pressure waveform analysis. This system offers several benefits such as sensitivity, convenience, and real-time application. It is used to assess volume status and enable optimal fluid management under positive pressure ventilation in high-risk surgical patients. Moreover, arterial pressure waveform analysis is superior to central venous pressure monitoring in terms of predicting volume responsiveness. Several studies have shown the benefits of SVV guidance during the intraoperative period in mechanically ventilated patients, including improved hemodynamic stability, decreased serum lactate levels, a lower incidence of postoperative complications, and shortened hospital stays. However, the reliability of arterial waveform analysis is influenced by certain conditions, such as tidal volume greater than 8 ml/kg, normal right ventricular function, absence of cardiac arrhythmias, and normal respiratory mechanics.

Perioperative fluid management is a crucial aspect of anesthesia for liver resection and is divided into two phases: the "fluid-restrictive" phase during parenchymal transection and the "resuscitative" phase after the completion of liver resection. In the first phase, intraoperative fluid administration can be restricted, and vasopressors may be administered to maintain hemodynamic stability. However, the optimal balance of fluid volumes and vasopressors is unclear. In the second phase, liberal fluid administration should be employed for resuscitation to reduce the risk of postoperative organ hypoperfusion, oliguria, and metabolic acidosis.

The utilization of stroke volume variation (SVV) for guiding fluid therapy in liver resection has been reported. Central venous pressure (CVP) monitoring was found to correlate significantly with SVV values during liver resection, demonstrating that a CVP of 3 mmHg correlated with an SVV of 13%, while a CVP of -1 to 1 mmHg corresponded to an SVV of 18-21%. Maintaining a high stroke volume variation of 10-20% as the target value during the restrictive phase has been shown to result in significantly lower amounts of intraoperative blood loss compared to patients maintained with a central venous pressure of less than 5 mmHg. Moreover, previous publications have shown that a high SVV (SVV 10-20%) compared to a low SVV (SVV <10%) reduces blood loss during liver resection. Additionally, goal-directed therapy (GDT) using the stroke volume variation parameter can guide the resuscitative phase during liver transection, potentially preventing excessive fluid administration after liver resection and helping to maintain a balanced fluid status postoperatively.

Objective

The purpose of this study is to compare the efficacy of maintaining high stroke volume variation versus low central venous pressure in minimizing perioperative blood loss during open liver resection. The primary and secondary objectives are as follows:

Primary Objective

To compare intraoperative blood loss between patients maintained with high stroke volume variation and those maintained with low central venous pressure during open liver resection by assessing:

* Blood loss during the liver transection phase
* Total blood loss Intraoperative blood loss will be estimated by combining the measured volume of suctioned blood and the measured weight of sponges and gauzes.

Secondary objectives To compare

1. Intraoperative transfusion

   * Intraoperative allogeneic packed red cell transfusion during the operation.
   * Intraoperative blood product transfusion during the operation.
2. Postoperative transfusion within 72 hours

   * Postoperative allogeneic packed red cell transfusion during admission, excluding the operating room.
   * Postoperative blood product transfusion during admission, excluding the operating room.
3. Surgical field bleeding

   - Classified by the same surgical team using the bleeding score of the hepatic surgical field.
4. Postoperative Major Complications

   - Identified and graded by the Clavien-Dindo classification.
5. Postoperative Acute Kidney Injury

   - Assessed and staged for severity according to Kidney Disease Improving Global Outcomes Outcomes (KDIGO) Clinical Practice Guidelines
6. Post-hepatectomy liver failure
7. Serum Lactate Level

   * Before liver resection
   * After completion of liver resection
   * After fluid resuscitation
8. Reoperation
9. Postoperative Length of Intensive Care Unit Stay
10. Postoperative Length of Hospital Stay
11. Postoperative In-Hospital Mortality
12. 30-Day Readmission
13. Postoperative 30-Days Mortality

ELIGIBILITY:
Inclusion Criteria:

* All genders, age 18 to 70 years old
* American Society of Anesthesiologists (ASA) physical status classification of I-III
* The patients who scheduled in elective open liver resection and diagnosed Hepatocellular Carcinoma, Cholangiocarcinoma, Liver metastasis, and Benign malignant tumor.

Exclusion Criteria:

* Pregnancy
* Active cardiac conditions (unstable coronary syndromes, decompensated heart failure, significant arrhythmias, severe valvular disease, active coronary artery disease within 6 months prior surgery)
* History of significant cerebrovascular disease (Patients with clinically significant stroke/CVA within 6 months prior surgery, severe carotid stenosis)
* Renal dysfunction (GFR < 60 ml/min/1.73 m²)
* Abnormal coagulation parameters (INR >1.5 not on warfarin and/or platelet count <100,000)
* Preoperative autologous blood donation
* Tumor size > 10 cm.
* Previous liver resection

Withdrawal criteria:

* Unresectable tumor
* Persistent intraoperative hypotension that cannot be corrected with vasopressors.
* Cardiac arrest during operation
* Low central venous pressure (CVP < 5 mmHg) or high stroke volume variation (SVV >13%) cannot be achieved before and during liver parenchymal transection.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2024-11-25 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Intraoperative blood loss during parenchymal transection phase and entire operation | From enrollment to the end of operation
  To compare intraoperative blood loss between patients maintained with high stroke volume variation and those maintained with low central venous pressure during open liver resection by assessing:
  * Blood loss during the liver transection phase
  * Total blood loss Intraoperative blood loss will be estimated by combining the measured volume of suctioned blood and the measured weight of sponges and gauzes.

SECONDARY OUTCOMES:
Allogenic blood transfusion and postoperative morbidity and mortality rate | From enrollment to the postoperative day 30
  Secondary objectives To compare
  1. Intraoperative transfusion
     * Intraoperative allogeneic packed red cell transfusion during the operation.
     * Intraoperative blood product transfusion during the operation.
  2. Postoperative transfusion within 72 hours
     * Postoperative allogeneic packed red cell transfusion during admission, excluding the operating room.
     * Postoperative blood product transfusion during admission, excluding the operating room.
  3. Surgical field bleeding
     - Classified by the same surgical team using the bleeding score of the hepatic surgical field.
  4. Postoperative Major Complications
     - Identified and graded by the Clavien-Dindo classification.
  5. Postoperative Acute Kidney Injury
     - Assessed and staged for severity according to Kidney Disease Improving Global Outcomes Outcomes (KDIGO) Clinical Practice Guidelines
  6. Post-hepatectomy liver failure
  7. Serum Lactate Level
     * Before liver resection
     * After completion of liver resection
     * After fluid resuscitation
  8. Reoperation

CONTACTS AND LOCATIONS:
Overall Officials: Warangkana Lapisatepun, MD. PhD., Principal Investigator — Chiang Mai University
Locations (1):
- Department of Anesthesiology, Faculty of Medicine, Chiang Mai University, Chiang Mai, Chiangmai, Thailand

IPD SHARING:
Plan to Share IPD: Yes
De-identified data from the study will be made available upon reasonable request to other researchers for further analysis and validation, in alignment with data sharing principles and participant confidentiality.

REFERENCES:
- [Result] Dunki-Jacobs EM, Philips P, Scoggins CR, McMasters KM, Martin RC 2nd. Stroke volume variation in hepatic resection: a replacement for standard central venous pressure monitoring. Ann Surg Oncol. 2014 Feb;21(2):473-8. doi: 10.1245/s10434-013-3323-9. Epub 2013 Oct 23. PMID 24150192